CLINICAL TRIAL: NCT01339065
Title: The Effect of Ketamine on Production of Inflammatory Markers in Post Operative Patients in Mulago Hospital: A Randomized Clinical Trial
Brief Title: The Effect of Ketamine on Production of Inflammatory Markers in Post Operative Patients in Mulago Hospital
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Responsible Party: Dr luggya Tonny Stone, Makerere University, College Of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: MUK CHS
Record Dates: First submitted 2011-04-19; First posted 2011-04-20 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Post Operative Inflammatory Marker Levels
Keywords: ketamine; inflammatory; pro inflammatory; pro inflammatory markers IL-6 and IL-1beta
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Active Comparator): will be given low sub-anesthetic doses of Ketamine 0.5mg/kg.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): will get placebo treatment
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — determining the effect of low dose sub anesthetic doze of ketamine and placaebo on post operative patients

SUMMARY:
. Null Hypothesis: Giving low doze ketamine (0.5mg/kg) given preoperatively to adult patients undergoing elective surgery, in Mulago hospital, will not have a reduction effect on the levels of IL-6 & IL-1β pro inflammatory markers by 48 hours.

. Alternate Hypothesis: Giving low doze ketamine (0.5mg/kg) given preoperatively to adult patients undergoing elective surgery, in Mulago hospital, will have a reduction effect on the levels of IL-6 & IL-1β pro inflammatory markers by 48 hours.

DETAILED DESCRIPTION:
RESEARCH QUESTION Can 0.5mg/kg of Ketamine given preoperatively have an effect on the levels of pro-inflammatory markers?

Primary specific Outcome: changes/deviations from baseline levels of IL- 6 pro-inflammatory markers of after surgery at PACU, 24 and 48 hours.

Secondary specific Outcome: changes/deviations from baseline levels of IL-1β pro-inflammatory markers of after surgery at PACU, 24 and 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Consented patients due for elective surgery
* Adult patients 18- 70 year old
* ASA I- ASA II scoring patients, who are normal patients or those with mild systemic illness

Exclusion Criteria:

* Emergency cases that will already have high levels of inflammatory markers secreted in their system by incision time e.g. road traffic accidents
* Patients with chronic / severe hypertension
* Febrile Patients (T >38°C)
* Persistently raised blood pressures above 140/90 for 2 consistent readings 15 minutes apart
* Patients with pheochromocytoma
* Spinal and local infiltration anaesthesia cases
* Neuro surgery patients whom Ketamine is contra indicated
* Epilepsy patients
* ASA IIIE and above
* Patients receiving Aspirin prophylaxis
* Chronic inflammatory disease states such as hyperparathyroidism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-05 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
changes/deviations from baseline levels of IL-6 pro-inflammatory markers of after surgery | 48 hours
  changes/deviations from baseline levels of IL-6 pro-inflammatory markers of after surgery at Post Anesthesia Care Unit, 24 and 48 hours

SECONDARY OUTCOMES:
changes/deviations from baseline levels of IL-1β pro-inflammatory markers of after surgery | 48 hours
  changes/deviations from baseline levels of IL-1β pro-inflammatory markers of after surgery at PACU, 24 and 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Mulago Hospital National Refferal, surgical wards, Kampala, Uganda

REFERENCES:
- [Derived] Luggya TS, Roche T, Ssemogerere L, Kintu A, Kasumba JM, Kwizera A, Tindimwebwa JV. Effect of low-dose ketamine on post-operative serum IL-6 production among elective surgical patients: a randomized clinical trial. Afr Health Sci. 2017 Jun;17(2):500-507. doi: 10.4314/ahs.v17i2.25. PMID 29062346